CLINICAL TRIAL: NCT06652399
Title: A Cohort Study: to Assess the Value of Cardiovascular Imaging in Pediatric Myocarditis
Brief Title: Cardiovascular Imaging in Pediatric Myocarditis
Status: Enrolling by invitation | Type: Observational
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Ling-Yi Wen, Principal Investigator, West China Second University Hospital
Other Study IDs: WestChinaSUH2023094
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Myocarditis
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the whole-blood sample will be collected for laboratory tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with pediatric myocarditis: Patients diagnosisd or suspected myocarditis based on the Diagnostic Recommendation for Myocarditis in Children (version 2018).

SUMMARY:
This study aims to utilize cardiac magnetic resonance (CMR) to assist in the clinical diagnosis, conduct consecutive assessments for myocardial tissue in pediatrics with myocarditis, and explore effective predictive factors for adverse outcomes in pediatric myocarditis.

Participants will undergo baseline collection, laboratory tests, echocardiography, and CMR. All the consecutive data will be used to analyze the association with the diagnosis and prognosis of pediatric myocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed or suspected pediatric myocarditis based on Diagnostic Recommendation for Myocarditis in Children (version 2018).
* Age between 1 to 18 years old.

Exclusion Criteria:

* Previous history of cardiovascular disease ( e.g. congenital heart disease, cardiomyopathy, rheumatic heart disease, valvular disease ).
* MRI examination contraindications ;
* Gadolinium contrast agent contraindications ;
* CT examination contraindications ;
* Comparison of iodine content.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: From the past to April 2032, pediatric patients diagnosed or suspected myocarditis were recruited from West China Second University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2032-11-01 (Estimated); Study Completion 2033-04-01 (Estimated)

PRIMARY OUTCOMES:
Adverse cardiovascular events | 10 years after the onset
  including all-cause death, orthotopic heart transplantation(HTx), malignant arrhythmia, readmission due to heart failure, progression to DCM.

SECONDARY OUTCOMES:
Secondary cardiovascular adverse events | 10 years after the onset
  including mild reduction of cardiac function, persistent mild AVB and other arrhythmias, left chest tightness, palpitations and other clinical symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferreira VM, Schulz-Menger J, Holmvang G, Kramer CM, Carbone I, Sechtem U, Kindermann I, Gutberlet M, Cooper LT, Liu P, Friedrich MG. Cardiovascular Magnetic Resonance in Nonischemic Myocardial Inflammation: Expert Recommendations. J Am Coll Cardiol. 2018 Dec 18;72(24):3158-3176. doi: 10.1016/j.jacc.2018.09.072. PMID 30545455
- [Background] Caforio AL, Pankuweit S, Arbustini E, Basso C, Gimeno-Blanes J, Felix SB, Fu M, Helio T, Heymans S, Jahns R, Klingel K, Linhart A, Maisch B, McKenna W, Mogensen J, Pinto YM, Ristic A, Schultheiss HP, Seggewiss H, Tavazzi L, Thiene G, Yilmaz A, Charron P, Elliott PM; European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Current state of knowledge on aetiology, diagnosis, management, and therapy of myocarditis: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 Sep;34(33):2636-48, 2648a-2648d. doi: 10.1093/eurheartj/eht210. Epub 2013 Jul 3. PMID 23824828
- [Background] Kantor PF, Lougheed J, Dancea A, McGillion M, Barbosa N, Chan C, Dillenburg R, Atallah J, Buchholz H, Chant-Gambacort C, Conway J, Gardin L, George K, Greenway S, Human DG, Jeewa A, Price JF, Ross RD, Roche SL, Ryerson L, Soni R, Wilson J, Wong K; Children's Heart Failure Study Group. Presentation, diagnosis, and medical management of heart failure in children: Canadian Cardiovascular Society guidelines. Can J Cardiol. 2013 Dec;29(12):1535-52. doi: 10.1016/j.cjca.2013.08.008. PMID 24267800
- [Background] JCS Joint Working Group. Guidelines for diagnosis and treatment of myocarditis (JCS 2009): digest version. Circ J. 2011;75(3):734-43. doi: 10.1253/circj.cj-88-0008. Epub 2011 Feb 4. No abstract available. PMID 21304213
- [Background] Howlett JG, McKelvie RS, Arnold JM, Costigan J, Dorian P, Ducharme A, Estrella-Holder E, Ezekowitz JA, Giannetti N, Haddad H, Heckman GA, Herd AM, Isaac D, Jong P, Kouz S, Liu P, Mann E, Moe GW, Tsuyuki RT, Ross HJ, White M; Canadian Cardiovascular Society. Canadian Cardiovascular Society Consensus Conference guidelines on heart failure, update 2009: diagnosis and management of right-sided heart failure, myocarditis, device therapy and recent important clinical trials. Can J Cardiol. 2009 Feb;25(2):85-105. doi: 10.1016/s0828-282x(09)70477-5. PMID 19214293